CLINICAL TRIAL: NCT05410119
Title: An 8-week Resilience-based Community Group Intervention Program for Parents Who Have Lost an Only Child in China
Brief Title: A Community-based Resilience Group Psychotherapy for Only-child Loss Parents in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Anni Wang, Lecturer, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resilience Group Psychotherapy
Record Dates: First submitted 2022-05-27; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience group (Experimental)
  Interventions: Behavioral: 8-week Resilience Group Psychotherapy
- Controlled group (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: 8-week Resilience Group Psychotherapy — Resilience Group Psychotherapy was intervened by a psychotherapy developed by the researchers. The resilience promotion therapy lasts 8 weeks, and also has a group intervention in each week. The themes of each week are start-up, mutual help, trust in yourself, thanksgiving feedback, care for yourself, emotional management, end-up.
  Arms: Resilience group
Other: Usual care — Usual care means treating as usual, such as regular home visit.
  Arms: Controlled group

SUMMARY:
Two communities in Changsha was selected, where principle investigators' institution located, to recruit 80 participants into intervention group and control group. Resilience therapy group was intervened by a psychotherapy developed by the researchers, which lasts 8 weeks. The themes of each week are start-up, mutual help, trust in yourself, thanksgiving feedback, care for yourself, emotional management, end-up. Measurement was conducted before the intervention, immediately after intervention, 3-month after intervention, and 12-month after intervention. A questionnaire was used during each measurement, including several scales in it, including resilience and depression.The saliva test of Dehydroepiandrosterone was also done in each measurement.

ELIGIBILITY:
Inclusion Criteria:

1. had only one child but now passed away;
2. failed to have another children;
3. volunteered to participate;
4. the score of resilience was under 72 points indicating a lower or middle level

Exclusion Criteria:

1. in the acute bereavement period (<6 months);
2. unable to participate in activities due to severe physical illness;
3. receiving drug treatment for mental illness;
4. receiving other psychological therapy

Min Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change of resilience | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention
  A kind of ability to bounce back from adversity measured by Connor-Davidson Resilience Scale, with higher score reflecting higher level of resilience, ranging from 0-100.
Change of depression | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention.
  Depressive mood in recent two weeks measured by Zung Self-rated Depression Scale, with higher score reflecting higher level of depression, ranging from 0-80.

SECONDARY OUTCOMES:
Change of subjective well-being | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention.
  A feeling of happiness measured by Campbell Index of well-being, with higher score reflecting higher subjective well-being, ranging from 1.1 to 14.7.
Change of social avoidance | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention.
  The phenomenon that a person is absent from normal social interaction with others measured by Social Avoidance and Distress Scale, with higher score reflecting higher social avoidance, ranging from 0 to 7.
Change of sleeping quality | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention.
  Sleep quality in recent month measured by Pittsburgh sleep quality index, with higher score reflecting bad quality, ranging from 0 to 23.
Change of post traumatic growth | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention.
  The positive growth after an adversity measured by Post Traumatic Growth Inventory, with higher score reflecting higher growth, ranging from 20 to 120.
Change of concentration of dehydroepiandrosterone in saliva | Change from before intervention, immediately after intervention,3-month after intervention, to 12-month after intervention.
  A kind of hormone that reflects the person's psychological stress collected by saliva collection tube by chewing the sterile cotton strips for 60 seconds, with higher concentration reflecting higher dehydroepiandrosterone level. The unit is pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT05410119/Prot_SAP_000.pdf